CLINICAL TRIAL: NCT04104477
Title: Carpometacarpal Osteoarthritis: Towards Identification of Biomechanical, Neuromuscular, and Somatosensory Mechanisms
Brief Title: Thumb Osteoarthritis: A Cross-Sectional Study of Mechanisms
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201900693-N; OCR20393 (Other: UF OnCore); KL2TR001429 (NIH)
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Carpometacarpal Osteoarthritis
Keywords: thumb, trapeziometacarpal, first metacarpal, trapezium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- End-Stage CMC OA: Individuals in this group had radiographic evidence of end-stage CMC OA defined as Eaton-Littler Stage III or Stage IV.
  During testing, participants will be asked to perform range of motion tasks, as well as strength tasks at varying effort levels (maximal and sub-maximal). Through a combination of quantitative testing and self-reported assessments, data on experimental pain, clinical pain, hand function, and disease severity will be reported.
  Interventions: Other: Range of Motion Tasks; Other: Strength Tasks
- Early-Stage CMC OA (Control): Individuals in this group had radiographic evidence of early-stage CMC OA defined as Eaton-Littler Stage I or Stage II. Note, the Eaton-Littler scale does not include a stage 0, thus no evidence of disease falls under Stage I.
  During testing, participants will be asked to perform range of motion tasks, as well as strength tasks at varying effort levels (maximal and sub-maximal). Through a combination of quantitative testing and self-reported assessments, data on experimental pain, clinical pain, hand function, and disease severity will be reported.
  Interventions: Other: Range of Motion Tasks; Other: Strength Tasks

INTERVENTIONS:
Other: Range of Motion Tasks — Participants will perform range of motion (thumb only) to evaluate fine and gross motor function.
Other: Strength Tasks — Participants will perform strength (pinch and grip) tests to evaluate fine and gross motor function.

SUMMARY:
This study examines carpometacarpal osteoarthritis (CMC OA) and aims to elucidate the biomechanical, neuromuscular, and somatosensory mechanisms that contribute to CMC OA symptoms by using orthopaedic biomechanics and quantitative pain testing. Completion of this study will provide a comprehensive dataset describing how movement strategies (muscle activity and joint posture) as well as experimental and clinical pain differ between individuals with CMC OA and age-matched controls.

DETAILED DESCRIPTION:
This study was funded by that National Institutes of Health through KL2 TR001429 and was registered as a clinical trial at the request of the funding agency. The goal of this exploratory, career development project was to conduct an observational, cross-sectional study of individuals with and without carpometacarpal osteoarthritis (CMC OA). Interestingly, even though approximately a third of postmenopausal women have radiographic evidence of CMC OA, less than ten percent of all women visit the doctor with painful symptoms. This disconnect between radiographic evidence of disease and presence of painful, clinical symptoms makes CMC OA challenging to study. Here, participants were recruited into two groups: CMC OA and age-matched controls. Participants with CMC OA were defined as those recruited from orthopaedic clinics with a diagnosis of CMC OA. Age-matched controls were defined as those recruited from the community who reported during screening that they had no pain or clinical symptoms of CMC OA. All participants participated in two sessions, a biomechanics session to evaluate movement (muscle activity, joint posture) and a somatosensory testing session to evaluate pain sensitization. All participants also completed clinical outcome measures and a hand x-ray. Analyses were completed on two groups based on radiographic evidence of CMC OA: early-stage and end-stage. Note, participant assignment to the analysis groups did not necessarily match the recruitment groups, as some control subjects had radiographic evidence of end-stage CMC OA and some individuals with diagnosed CMC OA had radiographic evidence of early-stage disease. The goal of this study was to build a small, comprehensive dataset describing how movement strategies (muscle activity and joint posture) as well as experimental and clinical pain differ across individuals with CMC OA.

ELIGIBILITY:
Inclusion Criteria:

* CMC OA Subjects:

  * female between the age of 40 to 90 years
  * end-stage CMC OA diagnosed by a board-certified clinician
* Age-Matched Control:

  * female between the age of 40 to 90 years
  * no joint or muscle pain in the hand or wrist

Exclusion Criteria:

* All Groups:

  * pregnant women; minors (under age 18); mentally disabled; any persons incarcerated, on parole, on probation, or awaiting trial
  * individuals with concomitant musculoskeletal pathologies (other than osteoarthritis) in the hand or wrist, including distal radius fracture, contracture, trigger finger, and carpal tunnel
  * individuals with history of uncontrolled diabetes, rheumatoid arthritis, muscular dysfunction, or neurological disease

Ages: 40 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All participants were recruited from North Central Florida. Participants with clinically-diagnosed CMC OA were recruited from local orthopaedic surgery clinics. Age-matched control subjects were recruited from the community.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Nichols, PhD, Principal Investigator — University of Florida
Locations (1):
- UF Health of University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Cohorts: Participants were recruited in two groups: CMC OA (diagnosed by clinician; recruited from orthopaedic clinic) and age-matched controls (recruited from community).
Pre-assignment Details: Analysis Cohorts: Using hand x-rays obtained during testing, participants were assigned to early-stage and end-stage OA cohorts for analysis. This accounted for the fact that individuals with CMC OA do not always seek clinical care.
Groups:
- End-Stage CMC OA; Early-Stage CMC OA (Control): During testing, participants will be asked to perform range of motion tasks, as well as strength tasks at varying effort levels (maximal and sub-maximal). Through a combination of quantitative testing and self-reported assessments, data on experimental pain, clinical pain, hand function, and disease severity will be reported.
  Range of Motion Tasks: Participants will perform range of motion (thumb only) to evaluate fine and gross motor function.
  Strength Tasks: Participants will perform strength (pinch and grip) tests to evaluate fine and gross motor function.
Period: Overall Study
Arm/Group | End-Stage CMC OA | Early-Stage CMC OA (Control)
Started | 15 | 16
Completed | 15 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | End-Stage CMC OA | Early-Stage CMC OA (Control) | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (10.4) | 59.9 (11.2) | 62.9 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 14 | 12 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 16 | 31
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.6 (4.6) | 26.8 (4.9) | 26.7 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Australian Canadian OA Hand Index (AUSCAN)
Description: The AUSCAN assesses health status and health outcomes in osteoarthritis of the hand. Participants complete 15 questions targeting their pain, stiffness, and physical function using a 5-point scale. The pain section is scored from 0-20, stiffness from 0-4, and function from 0-10. Higher score indicates worse self-reported outcomes.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | End-Stage CMC OA | Early-Stage CMC OA (Control)
Number analyzed (Participants) | 15 | 16
score on a scale
  AUSCAN Pain | 3.3 (2.6) | 1.3 (2.0)
  AUSCAN Stiffness | 2.0 (2.0) | 1.6 (2.3)
  AUSCAN Function | 3.7 (2.8) | 1.6 (2.2)

2. Primary Outcome: Disabilities of the Arm, Shoulder, and Hand (DASH)
Description: The DASH is a 30-item questionnaire that assesses an individual's ability to perform upper extremity activities. Participants rate the difficulty and interference of with daily life using a 5-point scale. Scores are reported from 0-100 with higher scores indicating worse self-reported outcomes.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | End-Stage CMC OA | Early-Stage CMC OA (Control)
Number analyzed (Participants) | 15 | 16
score on a scale | 27.8 (22.2) | 15.3 (16.4)

ADVERSE EVENTS:
Time Frame: Each participant completed three sessions, which could be completed in a single day or across multiple days. Sessions were typically scheduled within 1 to 2 weeks. Adverse event data was collected for each participant during the time period they were enrolled (i.e., during the three sessions), which typically did not exceed 1 month.
Description: Definitions based on interference with daily activities: Mild (easily tolerated, cause minimal discomfort), Moderate (sufficient discomfort to interfere with daily activities), Severe (prevents daily activities)
  Relationship to study: Unrelated (no association between study intervention and reported event), Related (definite causal relationship exists between the event and the study), Cannot be ruled out (the event might be related to the study, but could also be produced by other factors)
Arm/Group | End-Stage CMC OA | Early-Stage CMC OA (Control)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 1/15 | 1/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | End-Stage CMC OA (N=15) | Early-Stage CMC OA (Control) (N=16)
Vasovagal syncope (Nervous system disorders) | 1 (1) | 0 (0) — Vasovagal syncope in response to insertion of fine wire needle electrodes.
Imparied Vision (Eye disorders) | 0 (0) | 1 (1) — Impaired peripheral vision

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-05-29): https://cdn.clinicaltrials.gov/large-docs/77/NCT04104477/Prot_000.pdf
  • Informed Consent Form (2023-01-29): https://cdn.clinicaltrials.gov/large-docs/77/NCT04104477/ICF_001.pdf